CLINICAL TRIAL: NCT01137747
Title: A Phase I Trial of Carfilzomib in Adult Patients With Relapsed Acute Myeloid and Acute Lymphoblastic Leukemia
Brief Title: Carfilzomib in Patients With Relapsed Acute Myeloid or Acute Lymphoblastic Leukemia
Acronym: AML ALL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-0913 / 201107117
Record Dates: First submitted 2010-06-02; First posted 2010-06-04 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Leukemia
Keywords: carfilzomib; acute myeloid leukemia; acute lymphoblastic leukemia; phase I
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dose Level 0 (starting dose) (Experimental): Carfilzomib - 20 mg/m2 days 1 and 2, 27 mg/m2 for days 8 and 9 of cycle 1 only and, if days 8 and 9 are tolerated, may be increased to 36 mg/m2 for all subsequent doses. If DLT occurs while receiving 36 mg/m2, the dose may be reduced to 27 mg/m2.
  Dosing schedule is days 1, 2, 8, 9, 15, 16, 22, and 23 with no rest period during the 28 day cycle. Dose will be given IV over 30 minutes.
  2 cycles of treatment will be given. If the patient enters at leat a partial remission, then treatment may be extended up to 4 additional cycles.
  Interventions: Drug: Carfilzomib
- Dose Level +1 (Experimental): Carfilzomib - 20 mg/m2 days 1 and 2, 36 mg/m2 for days 8 and 9 of cycle 1 only and, if days 8 and 9 are tolerated, may be increased to 45 mg/m2 for all subsequent doses. If DLT occurs while receiving 45 mg/m2, the dose may be reduced to 36 mg/m2.
  Dosing schedule is days 1, 2, 8, 9, 15, 16, 22, and 23 with no rest period during the 28 day cycle. Dose will be given IV over 30 minutes.
  2 cycles of treatment will be given. If the patient enters at leat a partial remission, then treatment may be extended up to 4 additional cycles.
  Interventions: Drug: Carfilzomib
- Dose Level +2 (Experimental): Carfilzomib - 20 mg/m2 days 1 and 2, 45 mg/m2 for days 8 and 9 of cycle 1 only and, if days 8 and 9 are tolerated, may be increased to 56 mg/m2 for all subsequent doses. If DLT occurs while receiving 56 mg/m2, the dose may be reduced to 45 mg/m2.
  Dosing schedule is days 1, 2, 8, 9, 15, 16, 22, and 23 with no rest period during the 28 day cycle. Dose will be given IV over 30 minutes.
  2 cycles of treatment will be given. If the patient enters at leat a partial remission, then treatment may be extended up to 4 additional cycles.
  Interventions: Drug: Carfilzomib

INTERVENTIONS:
Drug: Carfilzomib
  Other Names: Kyprolis

SUMMARY:
This study is to test escalating doses of carfilzomib in patients with relapsed acute myeloid and acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
Several published studies have demonstrated the in vitro anti-leukemic activity of carfilzomib in leukemia cell lines as well as in primary human acute myeloid and acute lymphoblastic leukemia cells. The anti-leukemic activity of carfilzomib was consistently more potent than that of bortezomib, particularly at doses ≥27mg/m2. Importantly, patients treated on the phase I and phase II carfilzomib trials have had low rates of treatment-associated neuropathy. Several large collaborative groups have current phase II clinical trials that incorporate bortezomib into the treatment regimens for acute myeloid or acute lymphoblastic leukemia. Thus, there is a strong rationale for a study of carfilzomib, a potentially more potent proteasome inhibitor with less toxicity, in patients with relapsed acute leukemias.

ELIGIBILITY:
Inclusion Criteria:

Disease Related

* Relapsed acute myeloid leukemia or relapsed acute lymphoblastic leukemia. Patients with primary refractory AML or ALL (after standard induction chemotherapy) are also eligible if they have evidence of persistent disease documented by bone marrow biopsy done within 14 days of trial entry.
* Subjects must have disease documented on bone marrow biopsy done within 14 days of starting cycle 1

Demographic

* Males and females ≥ 18 years old.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.

Laboratory

* Peripheral blast count must be ≤ 30,000 on the first day of study drug administration. Leukopheresis and hydrea are acceptable measures of leuko-reduction prior to beginning the study drug.
* Adequate hepatic function with ALT/SGPT ≤ 2.5 x upper limit of normal (ULN) or ≤ 5.0 x ULN if the transaminase elevation is due to leukemic involvement. Serum bilirubin ≤ 2.0 x ULN.
* Adequate renal function with calculated creatinine clearance of ≥ 15 mL/min (calculated using the Cockcroft and Gault formula) or measured creatinine clearance ≥ 15 mL/min from 24 hour urine collection.
* Uric acid, if elevated, must be corrected to within laboratory normal range prior to dosing.

Ethical / Other

* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed.
* Women of childbearing age must have a negative serum pregnancy test within 7 days prior to initiating therapy and be willing to not become pregnant to by using effective contraception while undergoing treatment and for at least 3 months afterwards.
* Men must be willing not to father a new child while receiving therapy. They must use an effective barrier method of contraception during the study and for 3 months following the last dose.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria are not eligible to enroll in this study.

Disease Related

* Active CNS leukemia.
* Receiving any other investigational agents within 14 days of first dose of study drug.
* Had cytotoxic chemotherapy within 14 days of first dose of study drug. Leukopheresis and hydrea are allowed as specified per protocol
* Had allogeneic stem cell transplantation within 100 days of first dose of study drug. Patients with a history of graft-versus-host disease on a stable dose of immunosuppression and who are otherwise medically fit are eligible for the trial. Patients with active graft-versus host disease are excluded.
* Had radiotherapy within 14 days prior to study enrollment.
* Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis.

Concurrent Conditions

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, congestive heart failure of NYHA class 3 or 4, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements.
* Major surgery within three weeks before Day 1.
* Active hepatitis A, B, C infection.
* Known or suspected HIV infection or subjects who are HIV seropositive.
* Significant neuropathy (Grade 3, 4) at the time of study initiation.
* Patients in whom oral and/or IV fluid hydration is contraindicated, e.g., due to pre-existing pulmonary, cardiac, or renal impairment, will not be eligible to participate in the clinical trial.

Ethical / Other

-Female subjects who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-10; Primary Completion 2014-08 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) | End of cycle 1
  A hematologic adverse event will not be considered a dose-limiting toxicity. Tumor lysis syndrome is not a dose-limiting toxicity.

SECONDARY OUTCOMES:
To determine the rate of morphologic complete remission (CR) | Every 2 months for 2 years after first dose of study drug
To determine the rates of cytogenetic complete remission (CRc) morphologic complete remission with incomplete count recovery (CRi), overall response rate (CR+ CRi), partial remission (PR), stable disease and hematologic improvement. | Every 2 months for 2 years after first dose of study drug
To determine the time to response, remission duration, progression-free survival, event-free survival and overall survival of patients treated with carfilzomib. | Every 2 months for 2 years after first dose of study drug
To determine the safety and tolerability of carfilzomib by evaluating the number of participants with adverse events as a measure of safety and tolerability. | 30 days after end of treatment
To prospectively collect serum and bone marrow specimens to determine biomarkers of response and correlative ex vivo studies of the anti-leukemic activity of carfilzomib. | Baseline, Day 28 of cycles 1, 2, 4, 6 & End of Study

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Vij, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu